CLINICAL TRIAL: NCT05132517
Title: Relationship Between Magnesium Concentration in Blood and Kognitive Functions After Stroke
Brief Title: Magnesium and Cognition After Stroke
Status: Recruiting | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: MaSeKo
Record Dates: First submitted 2021-10-11; First posted 2021-11-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Cognition; Magnesium; Neurologic Disorder
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke Patients: Ischemic-/hemorragic stroke patients, who admitted on the stroke unit.
  Interventions: Diagnostic Test: Kölner Neuropsychologische Screening für Schlaganfall-Patienten

INTERVENTIONS:
Diagnostic Test: Kölner Neuropsychologische Screening für Schlaganfall-Patienten — The cognitive state of the patient is measure by the Kölner Neuropsychologische Screening (KöpSS) and by the Mini Mental Status Test (MMST). The MMST is a popular often used test, which makes comparisons to other international studies possible. However, even though this test was specifically designed for stroke patients, it has a limited sensibility. Thus the KöpSS is being used as an additional test demonstrating satisfactory sensibility and specificity. It is suitable for acute and subacute strokes and covers all stroke relevant domains.
  Other Names: KöpSS

SUMMARY:
Cognitive impairments such as memory impairments, word-finding difficulties, compromised orientation and perception are often observed in stroke patients.

Low serum-mg-concentrations are associated with cognitive impairments in ischemic stroke patients one month after stroke onset. It is not clear, if cognitive impairments after stroke is caused by the mg-deficiency or by the stroke itself. Until now, no studies investigating the relationship between mg-concentration, stroke severity and cognition during treatment course are available. Thus, this study aimed to investigate the relationship between mg-concentration and cognition of stroke patients.

DETAILED DESCRIPTION:
Stroke patients admitted to the stroke unit will be included. Initial mg-concentration in serum as well as stroke related measures (National Institutes of Health Stroke Scale, Scandinavian Stroke Scale, modified Rankin Scale) will be ealuated. Moreover, the cognitive abilities of the patient will be assessed within the first three days via the Kölner Neuropsychologische Screening for stroke patients as well as the Mini Mental Status Test.

During stroke rehabilitation mg-level, stroke related measures (NIHSS,SSS,MRS) as well as the cognitive tests (MMST,KöpSS) will be re-assed after 4 weeks, 3 month as well as at study end, which is defined as discharge from the clinic (death, transfer to another hospital without return after 4 weeks, discharge to long-term nursing/ home/hospice).

Attention-network of stroke patients are measeared if the patient undergo a MRi scan.

In this study following questions will be assessed:

1. What is the incidence of cognitive impairments in stroke patients?

   1. Are there differences between ischemic and hemorrhagic stroke patients?
   2. Are there age and/or gender differences?
2. Are there differences regarding the mg-concentration at admission in comparison to the follow-up (week 4 after admission, 3 month after admission) and between patients with/without cognitive impairments?
3. Is there a correlation between the mg-concentration and the stroke severity?
4. Is there a correlation between the scores of the different cognitive tests (MMST and KöpSS)?
5. Is there an association between the stroke severity, the cognitive impairments (KöpSS) and the neuronal attention network?

ELIGIBILITY:
Inclusion Criteria:

* ischemic/hemmorhagic stroke
* written consent form

Exclusion Criteria:

* pre-existing dementia or cognitive impairment before stroke onset
* pre-existing mental disorder (depression) or present/prior long-term treatment (> 6 months) with psychotropic drugs
* pre-existing malign tumor disease
* participation in another clinical trial within the past 30 days
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample is comprised of 80 stroke patients (ischemic/hemmorgic) of both genders and age ≥ 18 years. A written consent form is signed before inclusion.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum mg-concentration | day 1
  This study defines a reference value ranging from 1,8 to 2,53 mg/dl.
Change from Serum mg-concentration from admission at day 28 | day 28
  This study defines a reference value ranging from 1,8 to 2,53 mg/dl.
Change from Serum mg-concentration from admission at day 72 | day 72
  This study defines a reference value ranging from 1,8 to 2,53 mg/dl.
Change from Serum mg-concentration from admission at study end | up to 6 month
  This study defines a reference value ranging from 1,8 to 2,53 mg/dl.
Kölner Neuropsychologische Screening für Schlaganfall-Patienten (KöpSS) | day 3
  The score ranges from 0 to 108 points. If all subtest can be performed, a score <98 points identify an impaired cognition.
Change from Kölner Neuropsychologische Screening für Schlaganfall-Patienten (KöpSS) at day 28 | day 28
  The score ranges from 0 to 108 points. If all subtest can be performed, a score <98 points identify an impaired cognition.
Change from Kölner Neuropsychologische Screening für Schlaganfall-Patienten (KöpSS) at day 72 | day 72
  The score ranges from 0 to 108 points. If all subtest can be performed, a score <98 points identify an impaired cognition.
Change from Kölner Neuropsychologische Screening für Schlaganfall-Patienten (KöpSS) at study end | up to 6 month
  The score ranges from 0 to 108 points. If all subtest can be performed, a score <98 points identify an impaired cognition.
National Institutes of Health Stroke Scale | day 1
  0-5 points: mild stroke; 6-14 points: moderate stroke; 15- 24 points: severe stroke;
  ≥25 points: very severe stroke
Change from National Institutes of Health Stroke Scale at day 3 | day 3
  0-5 points: mild stroke; 6-14 points: moderate stroke; 15- 24 points: severe stroke;
  ≥25 points: very severe stroke
Change from National Institutes of Health Stroke Scale at day 28 | day 28
  0-5 points: mild stroke; 6-14 points: moderate stroke; 15- 24 points: severe stroke;
  ≥25 points: very severe stroke
Change from National Institutes of Health Stroke Scale at day 72 | day 72
  0-5 points: mild stroke; 6-14 points: moderate stroke; 15- 24 points: severe stroke;
  ≥25 points: very severe stroke
Change from National Institutes of Health Stroke Scale at study end | up to 6 month
  0-5 points: mild stroke; 6-14 points: moderate stroke; 15- 24 points: severe stroke;
  ≥25 points: very severe stroke
Lenght of stay | up to 6 month
  Lenght of stay will be assesse at discharge.

SECONDARY OUTCOMES:
Mini Mental State Test (MMST) | day 3
  30 - 28 points no dementia; 27 - 25 points mild cognitive decline; 24 - 18 points mild dementia; 17 - 10 points moderate dementia; < 10 points severe dementia
Change from Mini Mental State Test (MMST) at day 28 | day 28
  30 - 28 points no dementia; 27 - 25 points mild cognitive decline; 24 - 18 points mild dementia; 17 - 10 points moderate dementia; < 10 points severe dementia
Change from Mini Mental State Test (MMST) at day 72 | day 72
  30 - 28 points no dementia; 27 - 25 points mild cognitive decline; 24 - 18 points mild dementia; 17 - 10 points moderate dementia; < 10 points severe dementia
Change from Mini Mental State Test (MMST) at study end | up to 6 month
  30 - 28 points no dementia; 27 - 25 points mild cognitive decline; 24 - 18 points mild dementia; 17 - 10 points moderate dementia; < 10 points severe dementia
Modified Rankin Scale (MRS) | day 1
  0 - No symptoms;
  1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Change from Modified Rankin Scale (MRS) at day 3 | day 3
  0 - No symptoms;
  1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Change from Modified Rankin Scale (MRS) at day 28 | day 28
  0 - No symptoms;
  1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Change from Modified Rankin Scale (MRS) at day 72 | day 72
  0 - No symptoms;
  1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Change from Modified Rankin Scale (MRS) at study end | up to 6 month
  0 - No symptoms;
  1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Scandinavian Stroke Scale (SSS) | day 1
  Sum score range from 0 to 58 in the edited version,with 0 indicating severe neurological deficits and 58 indicating no neurological deficits.
Change from Scandinavian Stroke Scale (SSS) at day 3 | day 3
  Sum score range from 0 to 58 in the edited version,with 0 indicating severe neurological deficits and 58 indicating no neurological deficits.
Change from Scandinavian Stroke Scale (SSS) at day 28 | day 28
  Sum score range from 0 to 58 in the edited version,with 0 indicating severe neurological deficits and 58 indicating no neurological deficits.
Change from Scandinavian Stroke Scale (SSS) at day 72 | day 72
  Sum score range from 0 to 58 in the edited version,with 0 indicating severe neurological deficits and 58 indicating no neurological deficits.
Change from Scandinavian Stroke Scale (SSS) at study end | up to 6 month
  Sum score range from 0 to 58 in the edited version,with 0 indicating severe neurological deficits and 58 indicating no neurological deficits.
Early Rehabilitation Barthel Index (ERBI) | day 1
  Sum score range from -325 to 100 points,with 100 indicating independence in the activity of daily living.
Change from Early Rehabilitation Barthel Index (ERBI) at day 3 | day 3
  Sum score range from -325 to 100 points,with 100 indicating independence in the activity of daily living.
Change from Early Rehabilitation Barthel Index (ERBI) at day 28 | day 28
  Sum score range from -325 to 100 points,with 100 indicating independence in the activity of daily living.
Change from Early Rehabilitation Barthel Index (ERBI) at day 72 | day 72
  Sum score range from -325 to 100 points,with 100 indicating independence in the activity of daily living.
Change from Early Rehabilitation Barthel Index (ERBI) at study end | up to 6 month
  Sum score range from -325 to 100 points,with 100 indicating independence in the activity of daily living.
International Classification of Functioning Disability and Health (ICF) Assessment | day 1
  A core set consisting of 20 ICF items is used. The severity of each item is scored with zero ("no impairment") to four ("complete impairment").
Change from International Classification of Functioning Disability and Health (ICF) Assessment at day 28 | day 28
  A core set consisting of 20 ICF items is used. The severity of each item is scored with zero ("no impairment") to four ("complete impairment").
Change from International Classification of Functioning Disability and Health (ICF) Assessment at day 72 | day 72
  A core set consisting of 20 ICF items is used. The severity of each item is scored with zero ("no impairment") to four ("complete impairment").
Change from International Classification of Functioning Disability and Health (ICF) Assessment at study end | up to 6 month
  A core set consisting of 20 ICF items is used. The severity of each item is scored with zero ("no impairment") to four ("complete impairment").
Early Functional Abilities (EFA) | day 1
  Sum score range from 20 to 100 points,with 100 indicating no impairement.
Change from Early Functional Abilities (EFA) at day 28 | day 28
  Sum score range from 20 to 100 points,with 100 indicating no impairement.
Change from Early Functional Abilities (EFA) at day 72 | day 72
  Sum score range from 20 to 100 points,with 100 indicating no impairement.
Change from Early Functional Abilities (EFA) at study end | up to 6 month
  Sum score range from 20 to 100 points,with 100 indicating no impairement.
Adverse events and complications | up to 6 month
  All adverse events and complications will be documened.

OTHER OUTCOMES:
Demographics | day 1
  age, gender, ethnic origin
Location and size of insult | day 1
  evaluation by CCT or MRT (if available)
Charlson Comorbidity Index (CII) | day 1
  Charlson Comorbidity Index (CII) ranges from 0 to 42, which a score >5 points indicating a 85% mortality risk of one-year death.
Secondary diagnoses | day 1
  All secondary diagnoses (i.e. renal insufficiency, Diabetes mellitus, acidosis, alcohol use) which affects mg-absorption and/or -excretion are documented.
Medication | day 1
  Medication affecting mg-absorption and/or -excretion is documented.

CONTACTS AND LOCATIONS:
Overall Officials: Simone B Schmidt, Dr., Principal Investigator — BDH-Clinic Hessisch Oldendorf
Locations (1):
- Institute for Neurorehabilitation Research, BDH-Clinic Hessich Oldendorf, Hessisch Oldendorf, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tu X, Qiu H, Lin S, He W, Huang G, Zhang X, Wu Y, He J. Low levels of serum magnesium are associated with poststroke cognitive impairment in ischemic stroke patients. Neuropsychiatr Dis Treat. 2018 Nov 2;14:2947-2954. doi: 10.2147/NDT.S181948. eCollection 2018. PMID 30464479
- [Background] Kaesberg S, Fink GR, Kalbe E. [Neuropsychological assessment early after stroke--an overview of diagnostic instruments available in German and introduction of a new screening tool]. Fortschr Neurol Psychiatr. 2013 Sep;81(9):482-92. doi: 10.1055/s-0033-1350452. Epub 2013 Aug 28. German. PMID 23986457
- [Background] Classen und Nowitzki. Serum-Magnesium: Normalwerte und Referenzbereiche. Magnesium-Bulletin 1990; 12(4):127-132.